CLINICAL TRIAL: NCT01628237
Title: Effectiveness and Cost Management of Multicolumn Spinal Cord Stimulation in Neuropathic Pain Patients With Failed Back Surgery Syndrome
Acronym: ESTIMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-A011695-36
Record Dates: First submitted 2012-05-03; First posted 2012-06-26 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2014-03

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Monocolumn spinal cord stimulation (Active Comparator): Specify 5-6-5 Lead (only one column)
  Interventions: Device: comparison of spinal cord stimulation
- Multicolumn spinal cord stimulation (Experimental): Specify 5-6-5 Lead
  Interventions: Device: comparison of spinal cord stimulation

INTERVENTIONS:
Device: comparison of spinal cord stimulation
  Other Names: Specify(TM) 5-6-5 lead (Medtronic)

SUMMARY:
Failed back surgery syndrome (FBSS) constitutes a frequent pathology, generates a severe handicap for patients and represents a considerable expense for healthcare system. Neurostimulation has currently not been validated in the treatment of back pain because of technological limitations in implantable spinal cord stimulation (SCS). The lack of a validated technique for back pain relief has prompted the development of newer devices, including leads with increased number of contacts (up to 16) and various geometric arrangements, the objective of which is to cover a larger area while attempting to extend, steer, or focus the electric field of the stimulation within the spinal cord regions. This led companies to design a new generation of multicolumn surgical leads that allow the activation of longitudinal and transverse electric fields (multicolumn spinal cord stimulation, MSCS) in order to provide bilateral paresthesia coverage of back pain.

The objective of this study is to compare the analgesic efficacy of MSCS (using longitudinal and transverse electric stimulation) versus mono-column spinal cord stimulation (CSCS, using axial stimulation, actually represented by quadripolar or octopolar lead) on the treatment of lumbar pain.

A total of 115 patients will be randomized to either CSCS or MSCS. Patients, between 18 and 80 years old suffering from refractory neuropathic pain of radicular origin with associated back pain will be included. Patients will be divided into two groups. One group with MSCS during the 12 months after the new generation electrode implantation and one group with CSCS during 6 months and MSCS between 6 and 12 months after the new generation electrode implantation.

The following parameters will be evaluated during this study: overall pain VAS, leg pain VAS, back pain VAS, Oswestry disability index, Montgomery and Asberg Depression Rating scale, Brief Anxiety Scale and the Euro Quality of Life-5 Dimension Health questionnaire and costing in relation to surgery and patient management.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 80 years
* Presence of FBSS ≥ 3 months after one or several spine surgery
* Presence of back and leg pain with documented neuropathic component (DN4)
* Having failed well conducted conservative treatment
* Meeting the criteria for a test of spinal cord stimulation as recommended by HAS (multidisciplinary consultation, psychological evaluation
* Presence of uni-or bilateral radicular pain with severe intensity, VAS score greater than or equal to 50/100 (daily VAS mean on 5 consecutive days).
* Presence of associated back pain, as related to type "bar" or "tender points"
* Understanding and accepting the constraints of the study
* Covered by a French Health Insurance plan or benefiting of such as a third party in agreement with the French law (Huriet law n°88.1138 and modifications) on biomedical research
* Has given written consent to the study after receiving clear information.
* Absence of psychosis or evolutionary history of severe psychosis requiring hospitalization.
* Absence of progressive malignancy

Exclusion Criteria:

* Age < 18 and > 80 years
* Accessible because of back pain surgery 'mechanical' causal (discogenic back pain, spinal instability, spinal deformation)
* Presence of surgery, anesthetic and psychiatric contraindication for spinal cord stimulation system implantation
* Absence of informed consent signature
* Women of childbearing without effective contraception (hormonal / mechanical: oral, injectable, transdermal, implantable, intrauterine device or surgical: tubal ligation, hysterectomy, oophorectomy total) or breastfeeding.
* Subject not covered by a French Health Insurance plan or not benefiting of such as a third party
* Subject receiving enhanced protection: minors, pregnant women, nursing women, persons deprived of liberty by a judicial or administrative decision, adults under legal protection, and finally patients in emergency situations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogic Scale Low Back pain | Month 6

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital, Poitiers, France

REFERENCES:
- [Derived] Roulaud M, Durand-Zaleski I, Ingrand P, Serrie A, Diallo B, Peruzzi P, Hieu PD, Voirin J, Raoul S, Page P, Fontaine D, Lanteri-Minet M, Blond S, Buisset N, Cuny E, Cadenne M, Caire F, Ranoux D, Mertens P, Naous H, Simon E, Emery E, Gadan B, Regis J, Sol JC, Beraud G, Debiais F, Durand G, Guetarni Ging F, Prevost A, Brandet C, Monlezun O, Delmotte A, d'Houtaud S, Bataille B, Rigoard P. Multicolumn spinal cord stimulation for significant low back pain in failed back surgery syndrome: design of a national, multicentre, randomized, controlled health economics trial (ESTIMET Study). Neurochirurgie. 2015 Mar;61 Suppl 1:S109-16. doi: 10.1016/j.neuchi.2014.10.105. Epub 2014 Nov 20. PMID 25456442